CLINICAL TRIAL: NCT02528773
Title: Efficacy of ART to Interrupt HIV Transmission Networks
Acronym: ART-NET
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Susan Little, MD, Professor of Medicine, University of California, San Diego
Other Study IDs: 141105
Record Dates: First submitted 2015-05-13; First posted 2015-08-19 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Draws: Approximately 2 tablespoons (30 mL) of blood will be taken for blood tests and storage at each visit. Participants' blood will be tested for:
  * CD4+/CD8+ T-cell Count. This is a measure of the immune system; T-cells help the immune system fight infections.
  * HIV-1 RNA (Viral Load). This measures the amount of HIV in the blood.
  * HIV pol sequence. This measures the type of HIV in your blood.
  * Blood will be collected for storage for future HIV testing, studies to measure the amount of residual HIV that remains in people who are doing well on HIV treatment, genetic testing of the HIV virus and possible HLA genotype testing as determined by the results of this and future studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV positive: Persons newly diagnosed with HIV.

SUMMARY:
The investigators are conducting a study to learn more about the spread of HIV infection within different geographic regions and populations in San Diego County, with the goal of demonstrating that early use of HIV treatment can reduce the number of new infections in our community. At the study visits, participants will be examined by the study staff and asked to donate some blood. Participants will also be asked several questions about themselves, their background, behaviors, health, and the general geographic area in which they live. By collecting information about antiretroviral treatment choices that are made by study participants, the investigators will be better able to measure how effectively HIV treatment can interrupt (i.e., block) the spread of HIV. All of the information gathered at the study visits will be de-identified and analyzed. Study staff will use the information to better understand in which groups of people, and in what areas of San Diego, HIV is spreading most quickly. This information will be used to determine how well Antiretroviral Therapy (HIV treatment) by certain individuals can control the spread of HIV within the population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Newly diagnosed HIV infection
3. ART naïve (≤7 days ART, previous use of PEP or PrEP are not exclusions)
4. Subject must be able to provide written consent
5. Subject must agree to study specific specimen collections and visit schedule.
6. Subjects with newly diagnosed HIV infection who were identified on or after May 1, 2014 will be eligible for enrollment as long as they are co-enrolled to either AEH020 (project 08-0278) or AEH030 (project 140093) and DID meet the above study inclusion criteria (items at the time of enrollment to protocols AEH020 or AEH030).

Exclusion Criteria:

1. Any factor or factors that in the opinion of the local investigator that could prevent compliance with study requirements.
2. Contraindication to phlebotomy or specimen collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with newly diagnosed HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Network-level efficacy of ART as measured by the number of newly infected persons and network cluster growth over time | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Little, MD, Principal Investigator — UCSD
Locations (1):
- UCSD AntiViral Research Center, San Diego, California, United States

REFERENCES:
- See also: AntiViral Research Center website — http://avrc.ucsd.edu